CLINICAL TRIAL: NCT00031876
Title: Phase I/II Trial of Capecitabine With Weekly Paclitaxel for Advanced Breast Cancer
Brief Title: Capecitabine and Paclitaxel in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 26/00; EU-20135
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to determine the effectiveness of combining capecitabine and paclitaxel in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of capecitabine when combined with paclitaxel in patients with metastatic adenocarcinoma of the breast.
* Determine the clinical efficacy of the dose immediately preceding the MTD identified in phase I, in terms of response rate, time to treatment failure, time to disease progression, and overall survival, in these patients.
* Determine the toxicity of this regimen in these patients.
* Determine a well-tolerated drug combination for these patients.

OUTLINE: This is a dose-escalation, multicenter study of capecitabine.

Patients receive oral capecitabine twice daily on days 1-14 and paclitaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 or more of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the dose level immediately preceding the MTD.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for phase I and 15-46 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the breast
* Patients in phase I:

  * Evaluable disease
* Patients in phase II:

  * Bidimensionally measurable disease

    * Bone metastases are not considered measurable
* No known or clinically suspected CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 64

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC greater than 3,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2 times ULN (3 times ULN if liver metastases present)

Renal:

* Patients in phase I:

  * Creatinine clearance at least 50 mL/min
* Patients in phase I or II:

  * Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No grade 2 or greater atrioventricular block

Other:

* No cognitive impairment or severe psychiatric disorder
* No greater than grade 2 preexisting peripheral neuropathy
* No other prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* Able to tolerate steroid premedication

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* More than 6 months since prior adjuvant chemotherapy
* At least 1 year since prior continuous infusion of fluorouracil or capecitabine
* At least 1 year since prior taxane administered once every 3 weeks
* No prior taxane or capecitabine administered weekly
* No more than 1 prior chemotherapy regimen for metastatic or locally advanced breast cancer
* No other concurrent chemotherapy

Endocrine therapy:

* Prior hormonal treatment for metastatic breast cancer allowed
* No concurrent continuous glucocorticosteroids
* No concurrent systemic endocrine treatment for breast cancer

Radiotherapy:

* No concurrent radiotherapy to indicator lesion or more than 30% of bone marrow

Surgery:

* Not specified

Other:

* No other concurrent anticancer treatment
* No concurrent immunosuppressive drugs
* Concurrent bisphosphonates allowed if indicator lesion is non-bone
* Able to tolerate steroid premedication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2000-05; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Aebi, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Inselspital, Bern, Bern
  - UniversitaetsSpital, Zurich

REFERENCES:
- [Result] Gick U, Rochlitz C, Mingrone W, Pestalozzi B, Rauch D, Ballabeni P, Lanz D, Hess V, Aebi S. Efficacy and tolerability of capecitabine with weekly paclitaxel for patients with metastatic breast cancer: a phase II report of the SAKK. Oncology. 2006;71(1-2):54-60. doi: 10.1159/000100449. Epub 2007 Mar 5. PMID 17344671
- [Result] Uhlmann C, Ballabeni P, Rijken N, Brauchli P, Mingrone W, Rauch D, Pestalozzi BC, Rochlitz C, Aebi S; Swiss Group for Clinical Cancer Research; Swiss Institute for Applied Cancer Research. Capecitabine with weekly paclitaxel for advanced breast cancer: a phase I dose-finding trial. Oncology. 2004;67(2):117-22. doi: 10.1159/000080997. PMID 15539915